CLINICAL TRIAL: NCT01930188
Title: Efficacy and Safety of Semaglutide Once-weekly Versus Sitagliptin Once-daily as add-on to Metformin and/or TZD in Subjects With Type 2 Diabetes (SUSTAIN™ 2 - vs. DPP-4 Inhibitor)
Brief Title: Efficacy and Safety of Semaglutide Once-weekly Versus Sitagliptin Once-daily as add-on to Metformin and/or TZD in Subjects With Type 2 Diabetes
Acronym: SUSTAIN™ 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9535-3626; 2012-004827-19 (EudraCT Number); U1111-1135-8730 (Other: WHO); 132366 (Other: JapicCTI); CTRI/2014/05/004626 (Registry Identifier: Clinical Trial Registry India (CTRI))
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide; Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Semaglutide 0.5 mg + sitagliptin placebo (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Semaglutide 1.0 mg + sitagliptin placebo (Experimental)
  Interventions: Drug: semaglutide; Drug: placebo
- Sitagliptin 100 mg + semaglutide placebo 1.0 mg (Active Comparator)
  Interventions: Drug: sitagliptin; Drug: placebo
- Sitagliptin 100 mg + semaglutide placebo 0.5 mg (Active Comparator)
  Interventions: Drug: sitagliptin; Drug: placebo

INTERVENTIONS:
Drug: semaglutide — For subcutaneous injection (s.c., under the skin) once weekly. Will follow a fixed dose escalation regimen. The trial drug will be added on to the subject's stable pre-trial medication.
  Arms: Semaglutide 0.5 mg + sitagliptin placebo; Semaglutide 1.0 mg + sitagliptin placebo
Drug: sitagliptin — Tablets for oral administration once daily. The trial drug will be added on to the subject's stable pre-trial medication.
  Arms: Sitagliptin 100 mg + semaglutide placebo 0.5 mg; Sitagliptin 100 mg + semaglutide placebo 1.0 mg
Drug: placebo — Tablets for oral administration once daily. The trial drug will be added on to the subject's stable pre-trial medication.
  Arms: Semaglutide 0.5 mg + sitagliptin placebo; Semaglutide 1.0 mg + sitagliptin placebo
Drug: placebo — For subcutaneous injection (s.c., under the skin) once weekly. Will follow a fixed dose escalation regimen. The trial drug will be added on to the subject's stable pre-trial medication.
  Arms: Sitagliptin 100 mg + semaglutide placebo 0.5 mg; Sitagliptin 100 mg + semaglutide placebo 1.0 mg

SUMMARY:
This trial is conducted in Africa, Asia, Europe and South America. The aim of the trial is to evaluate efficacy and safety of semaglutide once-weekly versus sitagliptin once-daily as add-on to metformin and/or TZD (thiazolidinedione) in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Japan: Age minimum 20 years - Subjects diagnosed with type 2 diabetes and on stable treatment in a period of 90 days prior to screening with either metformin above or equal to 1500 mg (or maximum tolerated dose), pioglitazone above or equal to 30 mg (or maximum tolerated dose), rosiglitazone above or equal to 4 mg (or maximum tolerated dose) or a combination of either metformin/pioglitazone or metformin/rosiglitazone (doses as for individual therapies). Stable is defined as unchanged medication and unchanged dose - HbA1c 7.0 - 10.5 % (53 - 91 mmol/mol) (both inclusive) Exclusion Criteria: - Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using an adequate contraceptive method throughout the trial including the 5 weeks follow-up period (adequate contraceptive measures as required by local law or practice) - Any chronic disorder or severe disease which, in the opinion of the investigator, might jeopardise subject's safety or compliance with the protocol - Treatment with glucose lowering agent(s) other than stated in the inclusion criteria in a period of 90 days before screening. An exception is short-term treatment (below or equal to 7 days in total) with insulin in connection with inter-current illness - History of chronic or idiopathic acute pancreatitis - Screening calcitonin value above or equal to 50 ng/L (pg/mL) - Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN 2) - Impaired renal function defined as estimated glomerular filtration rate (eGFR) below 60 ml/min/1.73 m2 per modification of diet in renal disease (MDRD) formula (4 variable version) - Acute coronary or cerebrovascular event within 90 days before randomisation - Heart failure, New York Heart Association (NYHA) class IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1231 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2015-10-12 (Actual); Study Completion 2015-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (116):
- Argentina (3):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Mar del Plata
- Bulgaria (9):
  - Novo Nordisk Investigational Site, Burgas
  - Novo Nordisk Investigational Site, Haskovo
  - Novo Nordisk Investigational Site, Petrich
  - Novo Nordisk Investigational Site, Rousse
  - Novo Nordisk Investigational Site, Sliven
  - Novo Nordisk Investigational Site, Smolyan
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Stara Zagora
  - Novo Nordisk Investigational Site, Vratsa
- Czechia (5):
  - Novo Nordisk Investigational Site, Chrudim
  - Novo Nordisk Investigational Site, Ostrava
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Praha 4- Chodov
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Szeged
  - Novo Nordisk Investigational Site, Szombathely
- India (15):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Trivandrum, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Ludhiana, Punjab
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, New Delhi
- Japan (12):
  - Novo Nordisk Investigational Site, Asahikawa-shi, Hokkaido
  - Novo Nordisk Investigational Site, Ibaraki
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Kitakyushu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Mitaka-shi, Tokyo
  - Novo Nordisk Investigational Site, Mito-shi, Ibaraki
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Okayama-shi, Okayama
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Tokyo
- Mexico (4):
  - Novo Nordisk Investigational Site, Pachuca, Hidalgo
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
  - Novo Nordisk Investigational Site, Aguascalientes
- Norway (5):
  - Novo Nordisk Investigational Site, Ålesund
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Kløfta
  - Novo Nordisk Investigational Site, Kongsvinger
  - Novo Nordisk Investigational Site, Stavanger
- Portugal (7):
  - Novo Nordisk Investigational Site, Almada
  - Novo Nordisk Investigational Site, Coimbra
  - Novo Nordisk Investigational Site, Lisbon
  - Novo Nordisk Investigational Site, Matosinhos Municipality
  - Novo Nordisk Investigational Site, Tomar
  - Novo Nordisk Investigational Site, Viana do Castelo
  - Novo Nordisk Investigational Site, Vila Nova de Gaia
- Romania (4):
  - Novo Nordisk Investigational Site, Baia Mare, Maramureş
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
  - Novo Nordisk Investigational Site, Brasov
  - Novo Nordisk Investigational Site, Bucharest
- Russia (14):
  - Novo Nordisk Investigational Site, Barnaul
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Nizhny Novgorod
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Smolensk
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Tyumen
  - Novo Nordisk Investigational Site, Ufa
  - Novo Nordisk Investigational Site, Volgograd
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Yaroslavl
- South Africa (6):
  - Novo Nordisk Investigational Site, East London, Eastern Cape
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Krugersdorp, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- Spain (7):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Centelles (Barcelona)
  - Novo Nordisk Investigational Site, La Roca Del Vallés
  - Novo Nordisk Investigational Site, Lleida
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Seville
- Sweden (4):
  - Novo Nordisk Investigational Site, Kristianstad
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
- Thailand (3):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Bangkoknoi, Bangkok
  - Novo Nordisk Investigational Site, Nakhon Ratchasima
- Turkey (Türkiye) (7):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Çorum
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Konya
  - Novo Nordisk Investigational Site, Rize
  - Novo Nordisk Investigational Site, Trabzon
- Ukraine (6):
  - Novo Nordisk Investigational Site, Cherkasy
  - Novo Nordisk Investigational Site, Ivano-Frankivsk
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Odesa
  - Novo Nordisk Investigational Site, Vinnytsia
  - Novo Nordisk Investigational Site, Zaporizhia

REFERENCES:
- [Background] Fonseca VA, Capehorn MS, Garg SK, Jodar Gimeno E, Hansen OH, Holst AG, Nayak G, Seufert J. Reductions in Insulin Resistance are Mediated Primarily via Weight Loss in Subjects With Type 2 Diabetes on Semaglutide. J Clin Endocrinol Metab. 2019 Sep 1;104(9):4078-4086. doi: 10.1210/jc.2018-02685. PMID 30938762
- [Background] Rodbard HW, Bellary S, Hramiak I, Seino Y, Silver R, Damgaard LH, Nayak G, Zacho J, Aroda VR. GREATER COMBINED REDUCTIONS IN HbA1C >/=1.0% AND WEIGHT >/=5.0% WITH SEMAGLUTIDE VERSUS COMPARATORS IN TYPE 2 DIABETES. Endocr Pract. 2019 Jun;25(6):589-597. doi: 10.4158/EP-2018-0444. Epub 2019 Mar 13. PMID 30865526
- [Result] Ahrén B, Comas LM, Kumar H, Sargin M, Derving Karsbøl J, Jacobsen SH, Chow F. Efficacy and Safety of Once-weekly Semaglutide vs Sitagliptin as add-on to Metformin and/or Thiazolidinediones After 56 Weeks in Subjects With Type 2 Diabetes (SUSTAIN 2). Oral Presentation 12 Jun 2016 at American Diabetes Association - 76th Annual Scientific Sessions.
- [Result] Ahrén B, Masmiquel L, Kumar H, Sargin M, Derving Karsbøl J, Jacobsen SH, Chow F. Efficacy and Safety of Once-weekly Semaglutide vs Sitagliptin as add-on to Metformin and/or Thiazolidinediones After 56 Weeks in Subjects With Type 2 Diabetes (SUSTAIN 2). ePoster #767 presented 12 Sep 2016 at European Association for the Study of Diabetes - 52nd Annual Meeting.
- [Result] Ahren B, Masmiquel L, Kumar H, Sargin M, Karsbol JD, Jacobsen SH, Chow F. Efficacy and safety of once-weekly semaglutide versus once-daily sitagliptin as an add-on to metformin, thiazolidinediones, or both, in patients with type 2 diabetes (SUSTAIN 2): a 56-week, double-blind, phase 3a, randomised trial. Lancet Diabetes Endocrinol. 2017 May;5(5):341-354. doi: 10.1016/S2213-8587(17)30092-X. Epub 2017 Apr 3. PMID 28385659
- [Result] Petri KCC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Exposure-response analysis for evaluation of semaglutide dose levels in type 2 diabetes. Diabetes Obes Metab. 2018 Sep;20(9):2238-2245. doi: 10.1111/dom.13358. Epub 2018 Jun 15. PMID 29748996
- [Result] Ahren B, Atkin SL, Charpentier G, Warren ML, Wilding JPH, Birch S, Holst AG, Leiter LA. Semaglutide induces weight loss in subjects with type 2 diabetes regardless of baseline BMI or gastrointestinal adverse events in the SUSTAIN 1 to 5 trials. Diabetes Obes Metab. 2018 Sep;20(9):2210-2219. doi: 10.1111/dom.13353. Epub 2018 Jun 12. PMID 29766634
- [Result] Sharma R, Wilkinson L, Vrazic H, Popoff E, Lopes S, Kanters S, Druyts E. Comparative efficacy of once-weekly semaglutide and SGLT-2 inhibitors in type 2 diabetic patients inadequately controlled with metformin monotherapy: a systematic literature review and network meta-analysis. Curr Med Res Opin. 2018 Sep;34(9):1595-1603. doi: 10.1080/03007995.2018.1476332. Epub 2018 May 29. PMID 29764222
- [Result] DeVries JH, Desouza C, Bellary S, Unger J, Hansen OKH, Zacho J, Woo V. Achieving glycaemic control without weight gain, hypoglycaemia, or gastrointestinal adverse events in type 2 diabetes in the SUSTAIN clinical trial programme. Diabetes Obes Metab. 2018 Oct;20(10):2426-2434. doi: 10.1111/dom.13396. Epub 2018 Jul 9. PMID 29862621
- [Result] Carlsson Petri KC, Ingwersen SH, Flint A, Zacho J, Overgaard RV. Semaglutide s.c. Once-Weekly in Type 2 Diabetes: A Population Pharmacokinetic Analysis. Diabetes Ther. 2018 Aug;9(4):1533-1547. doi: 10.1007/s13300-018-0458-5. Epub 2018 Jun 15. PMID 29907893
- [Result] Aroda VR, Ahmann A, Cariou B, Chow F, Davies MJ, Jodar E, Mehta R, Woo V, Lingvay I. Comparative efficacy, safety, and cardiovascular outcomes with once-weekly subcutaneous semaglutide in the treatment of type 2 diabetes: Insights from the SUSTAIN 1-7 trials. Diabetes Metab. 2019 Oct;45(5):409-418. doi: 10.1016/j.diabet.2018.12.001. Epub 2019 Jan 4. PMID 30615985
- [Derived] Pulleyblank R, Larsen NB. Cost-Effectiveness of Semaglutide vs. Empagliflozin, Canagliflozin, and Sitagliptin for Treatment of Patients with Type 2 Diabetes in Denmark: A Decision-Analytic Modelling Study. Pharmacoecon Open. 2023 Jul;7(4):579-591. doi: 10.1007/s41669-023-00416-z. Epub 2023 May 13. PMID 37178435
- [Derived] Husain M, Bain SC, Holst AG, Mark T, Rasmussen S, Lingvay I. Effects of semaglutide on risk of cardiovascular events across a continuum of cardiovascular risk: combined post hoc analysis of the SUSTAIN and PIONEER trials. Cardiovasc Diabetol. 2020 Sep 30;19(1):156. doi: 10.1186/s12933-020-01106-4. PMID 32998732
- [Derived] Lingvay I, Capehorn MS, Catarig AM, Johansen P, Lawson J, Sandberg A, Shaw R, Paine A. Efficacy of Once-Weekly Semaglutide vs Empagliflozin Added to Metformin in Type 2 Diabetes: Patient-Level Meta-analysis. J Clin Endocrinol Metab. 2020 Dec 1;105(12):e4593-604. doi: 10.1210/clinem/dgaa577. PMID 32827435
- [Derived] Capehorn M, Ghani Y, Hindsberger C, Johansen P, Jodar E. Once-Weekly Semaglutide Reduces HbA1c and Body Weight in Patients with Type 2 Diabetes Regardless of Background Common OAD: a Subgroup Analysis from SUSTAIN 2-4 and 10. Diabetes Ther. 2020 May;11(5):1061-1075. doi: 10.1007/s13300-020-00796-z. Epub 2020 Mar 19. PMID 32193837
- [Derived] Husain M, Bain SC, Jeppesen OK, Lingvay I, Sorrig R, Treppendahl MB, Vilsboll T. Semaglutide (SUSTAIN and PIONEER) reduces cardiovascular events in type 2 diabetes across varying cardiovascular risk. Diabetes Obes Metab. 2020 Mar;22(3):442-451. doi: 10.1111/dom.13955. Epub 2020 Feb 5. PMID 31903692
- [Derived] DeSouza C, Cariou B, Garg S, Lausvig N, Navarria A, Fonseca V. Efficacy and Safety of Semaglutide for Type 2 Diabetes by Race and Ethnicity: A Post Hoc Analysis of the SUSTAIN Trials. J Clin Endocrinol Metab. 2020 Feb 1;105(2):dgz072. doi: 10.1210/clinem/dgz072. PMID 31769496
- [Derived] Jendle J, Birkenfeld AL, Polonsky WH, Silver R, Uusinarkaus K, Hansen T, Hakan-Bloch J, Tadayon S, Davies MJ. Improved treatment satisfaction in patients with type 2 diabetes treated with once-weekly semaglutide in the SUSTAIN trials. Diabetes Obes Metab. 2019 Oct;21(10):2315-2326. doi: 10.1111/dom.13816. Epub 2019 Jul 12. PMID 31215727
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 124 sites in 18 countries: Argentina: 4; Bulgaria: 10; Czech Republic: 5; Hong Kong: 1; Hungary: 4; India: 11; Japan: 14; Mexico: 5 Norway: 5; Portugal: 6; Romania: 5; Russian Federation: 17; South Africa: 7; Spain: 7: Sweden: 4; Thailand: 4; Turkey: 9; and Ukraine: 6 sites.
Groups:
- Semaglutide 0.5 mg + Sitagliptin Placebo: Semaglutide 0.5 mg administered subcutaneously (s.c., under the skin) once weekly, in the thigh, abdomen, or upper arm, at any time of day irrespective of meals. Sitagliptin placebo (0 mg) administered orally once daily.
- Semaglutide 1.0 mg + Sitagliptin Placebo: Semaglutide 1.0 mg administered subcutaneously (s.c., under the skin) once weekly, in the thigh, abdomen, or upper arm, at any time of day irrespective of meals. Sitagliptin placebo (0 mg) administered orally once daily.
- Sitagliptin + Semaglutide Placebo: Subjects were randomised to 2 different placebo arms (sitagliptin + semaglutide placebo 0.5 mg and sitagliptin + semaglutide placebo 1.0 mg). Both arms were pooled together for data analysis. Semaglutide placebo administered subcutaneously (s.c., under the skin) once weekly, in the thigh, abdomen, or upper arm, at any time of day irrespective of meals. Sitagliptin (100 mg) administered orally once daily.
Period: Overall Study
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo
Started | 409 | 409 | 407
Premature Discontinuation of Treatment | 53 (Subjects prematurely discontinued treatment were allowed to continue participation in the trial.) | 61 (Subjects prematurely discontinued treatment were allowed to continue participation in the trial.) | 32 (Subjects prematurely discontinued treatment were allowed to continue participation in the trial.)
Completed | 387 | 388 | 388
Not Completed | 22 | 21 | 19
Not completed — unclassified | 4 | 5 | 3
Not completed — Missing follow-up information | 2 | 2 | 3
Not completed — Lost to Follow-up | 5 | 2 | 2
Not completed — Death | 2 | 1 | 3
Not completed — Withdrawal by Subject | 9 | 11 | 8

BASELINE CHARACTERISTICS:
Population: Of 1231 randomised subjects, 6 were excluded: 1 subject each in the semaglutide 0.5 mg and 1.0 mg arms and 4 subjects in the sitagliptin arm were not exposed to trial treatment. Baseline characteristics were presented for 1225 subjects (Full Analysis Set), who received at least one dose of randomised semaglutide or sitagliptin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo | Total
Number analyzed (Participants) | 409 | 409 | 407 | 1225
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.2) | 56.0 (9.4) | 54.6 (10.4) | 55.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 204 | 199 | 605
  Male | 207 | 205 | 208 | 620
HbA1c [Mean (Standard Deviation); unit: percentage] | 8.01 (0.92) | 8.04 (0.93) | 8.17 (0.92) | 8.07 (0.93)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 89.93 (20.39) | 89.21 (20.74) | 89.29 (19.67) | 89.48 (20.26)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mmol/L] | 9.33 (2.38) | 9.29 (2.22) | 9.60 (2.16) | 9.40 (2.26)
Diastolic and Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Diastolic Blood pressure | 80.63 (9.76) | 80.87 (9.08) | 80.48 (8.70) | 80.66 (9.19)
  Systolic Blood pressure | 132.73 (16.09) | 132.56 (13.93) | 132.66 (14.58) | 132.65 (14.88)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin) From Baseline
Description: Change in HbA1c from baseline until week 56.Full analysis set (FAS=1225) included all randomised subjects who had received at least one dose of randomised semaglutide or sitagliptin.
Time Frame: Week 0, week 56
Population: Missing data imputed from a mixed model for repeated measurements for treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated haemoglobin
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo
Number analyzed (Participants) | 409 | 409 | 407
percentage of glycosylated haemoglobin | -1.32 (0.05) | -1.61 (0.05) | -0.55 (0.05)
Statistical Analysis 1: Comparison: Semaglutide 1.0 mg + Sitagliptin Placebo vs Sitagliptin + Semaglutide Placebo; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the upper limit of the two-sided 95% confidence interval for the estimated treatment difference between semaglutide 1.0 mg and sitagliptin was below the pre-specified non-inferiority margin (0.3 %); p < 0.0001, Mixed Models Analysis; Post-baseline responses analysed with mixed model for repeated measurements-treatment & country (fixed) & baseline (covariate) all nested within visit; treatment difference = -1.06, 95% CI 2-sided [-1.21 to -0.91]
Statistical Analysis 2: Comparison: Semaglutide 0.5 mg + Sitagliptin Placebo vs Sitagliptin + Semaglutide Placebo; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded if the upper limit of the two-sided 95% confidence interval for the estimated treatment difference between semaglutide 0.5 mg and sitagliptin was below the pre-specified non-inferiority margin (0.3 %); p < 0.0001, Mixed Models Analysis; Analysis done with mixed model for repeated measurements (treatment & country as fixed factors & baseline value as covariate) all nested within visit; treatment difference = -0.92, 95% CI 2-sided [-1.21 to -0.62]

2. Secondary Outcome: Change in Body Weight From Baseline
Description: Change in body weight from baseline to week 56. Full analysis set (FAS=1225) included all randomised subjects who had received at least one dose of semaglutide or sitagliptin.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo
Number analyzed (Participants) | 409 | 409 | 407
kilograms | -4.28 (0.25) | -6.13 (0.25) | -1.93 (0.26)

3. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline
Description: Change in fasting plasma glucose from baseline to week 56. Full analysis set (FAS=1225) included all randomised subjects who had received at least one dose of semaglutide or sitagliptin.
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo
Number analyzed (Participants) | 409 | 409 | 407
mg/dL | -37.38 (1.79) | -46.72 (1.78) | -19.85 (1.88)

4. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure From Baseline
Description: Change in systolic and diastolic blood pressure from baseline to week 56. Full analysis set (FAS=1225) included all randomised subjects who had received at least one dose of semaglutide or sitagliptin
Time Frame: Week 0, week 56
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo
Number analyzed (Participants) | 409 | 409 | 407
mmHg
  Systolic blood pressure | -5.07 (0.64) | -5.61 (0.63) | -2.29 (0.67)
  Diastolic blood pressure | -2.01 (0.42) | -1.91 (0.42) | -1.11 (0.44)

5. Secondary Outcome: Change in Patient Reported Outcome (PRO) Questionnaire Diabetes Treatment Satisfaction Questionnaire Status (DTSQs) From Baseline
Description: Full analysis set (FAS=1225) included all randomised subjects who had received at least one dose of semaglutide or sitagliptin. The DTSQs questionnaire was used to assess subjects' treatment satisfaction. This questionnaire contained 8 components and evaluates the diabetes treatment (including insulin, tablets and/or diet) in terms of convenience, flexibility and general feelings towards the treatment. The result presented is the 'Treatment Satisfaction' summary score, which is the sum of 6 of the 8 items of the DTSQs questionnaire. Response options range from 6 (best case) to 0 (worst case). Total scores for treatment satisfaction range from 0-36. Higher scores indicate higher satisfaction.
Time Frame: Week 0, week 56
Population: Out of the 1225 subjects in FAS, 76 in semaglutide 0.5 mg arm, 76 in semaglutide 1.0 mg arm, and 113 in placebo arm had missing data for the endpoint. Missing data imputed from a mixed model for repeated measurements for treatment and country as fixed factors and baseline value as covariate, all nested within visit.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo
Number analyzed (Participants) | 333 | 333 | 294
Units on a scale | 5.28 (0.23) | 5.91 (0.23) | 4.45 (0.24)

6. Secondary Outcome: Subjects Who Achieved HbA1c Below or Equal to 6.5% (48 mmol/Mol) American Association of Clinical Endocrinologists (AACE) Target (Yes/no)
Description: Subjects who achieved HbA1c ≤6.5% (48 mmol/mol) American Association of Clinical Endocrinologists (AACE) target (yes/no) after week 56 weeks of treatment.
Time Frame: After 56 weeks treatment
Population: Full analysis set (FAS=1225) included all randomised subjects who had received at least one dose of semaglutide or sitagliptin
Measure: Number; unit: Subjects
Arm/Group | Semaglutide 0.5 mg + Sitagliptin Placebo | Semaglutide 1.0 mg + Sitagliptin Placebo | Sitagliptin + Semaglutide Placebo
Number analyzed (Participants) | 409 | 409 | 407
Subjects
  Yes | 215 | 270 | 83
  No | 194 | 139 | 324

ADVERSE EVENTS:
Time Frame: Adverse events are reported for on-treatment period i.e from the date of initiation of trial product to the end of the on-treatment period (up to 56 weeks).
Description: Safety analysis set included all subjects exposed to at least one dose of semaglutide or sitagliptin. Number of deaths causally related to treatment is the data considered to present under 'total number of deaths resulting from adverse events'.
Groups:
- Semaglutide 1.0 mg + Sitagliptin Placebo: Semaglutide 1.0 mg once-weekly + Sitagliptin placebo once-daily
- Semaglutide 0.5 mg + Sitagliptin Placebo: Semaglutide 0.5 mg once-weekly + Sitagliptin placebo once-daily
- Sitagliptin 100 mg + Semaglutide Placebo 1.0 mg: Sitagliptin 100 mg once-daily + Semaglutide placebo 1.0 mg once-weekly
- Sitagliptin 100 mg + Semaglutide Placebo 0.5 mg: Sitagliptin 100 mg once-daily + Semaglutide placebo 0.5 mg once-weekly
Arm/Group | Semaglutide 1.0 mg + Sitagliptin Placebo | Semaglutide 0.5 mg + Sitagliptin Placebo | Sitagliptin 100 mg + Semaglutide Placebo 1.0 mg | Sitagliptin 100 mg + Semaglutide Placebo 0.5 mg
Serious Adverse Events (participants affected / at risk) | 30/409 | 30/409 | 13/204 | 16/203
Other Adverse Events (participants affected / at risk) | 197/409 | 208/409 | 75/204 | 85/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg + Sitagliptin Placebo (N=409) | Semaglutide 0.5 mg + Sitagliptin Placebo (N=409) | Sitagliptin 100 mg + Semaglutide Placebo 1.0 mg (N=204) | Sitagliptin 100 mg + Semaglutide Placebo 0.5 mg (N=203)
Abdominal lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of eyelid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gas poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoid operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Ketonuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligamentitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meniscus operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papilla of Vater stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Splenic lesion (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xanthelasma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 1.0 mg + Sitagliptin Placebo (N=409) | Semaglutide 0.5 mg + Sitagliptin Placebo (N=409) | Sitagliptin 100 mg + Semaglutide Placebo 1.0 mg (N=204) | Sitagliptin 100 mg + Semaglutide Placebo 0.5 mg (N=203)
Constipation (Gastrointestinal disorders) | 23 (29) | 18 (20) | 5 (5) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 27 (29) | 26 (28) | 6 (6) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 53 (85) | 53 (91) | 13 (17) | 16 (18)
Dyspepsia (Gastrointestinal disorders) | 20 (27) | 26 (28) | 4 (4) | 5 (7)
Headache (Nervous system disorders) | 29 (42) | 26 (81) | 9 (19) | 8 (10)
Influenza (Infections and infestations) | 22 (25) | 18 (23) | 13 (14) | 14 (16)
Lipase increased (Investigations) | 32 (38) | 33 (41) | 13 (16) | 16 (17)
Nasopharyngitis (Infections and infestations) | 29 (33) | 50 (63) | 19 (20) | 23 (31)
Nausea (Gastrointestinal disorders) | 72 (140) | 73 (110) | 13 (15) | 17 (23)
Pharyngitis (Infections and infestations) | 10 (12) | 7 (7) | 5 (5) | 13 (16)
Vomiting (Gastrointestinal disorders) | 41 (119) | 33 (49) | 6 (7) | 5 (9)

LIMITATIONS AND CAVEATS:
None reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigators(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.